CLINICAL TRIAL: NCT03637023
Title: Clinical and Rest-fMRI Effects of Virtual Reality Practice on Motor and Cognitive Symptoms in Parkinson's Disease, a Randomized Control Trial
Brief Title: Virtual Reality for Parkinson's Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: due to COVID-19 outbreak
Sponsor: Farzin Hajebrahimi, PT, MSc (Other)
Responsible Party: Sponsor-Investigator, Farzin Hajebrahimi, PT, MSc, Principle Investigator, Istanbul Medipol University Hospital
Organization: Istanbul Medipol University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PD-VR-2018
Record Dates: First submitted 2018-08-10; First posted 2018-08-17 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Parkinson Disease; Virtual Reality Therapy; Functional Magnetic Resonance Imaging
Keywords: fMRI; Virtual Reality Therapy; Exercise Therapy
MeSH Terms: conditions — Parkinson Disease | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (Experimental): Virtual Reality will be applied in addition to the Anti-parkinsonian medication given by the Neurologist.
  Interventions: Behavioral: Virtual Reality
- Exercise Therapy (Active Comparator): Exercise Therapy will be applied in addition to the Anti-parkinsonian medication given by the Neurologist.
  Interventions: Behavioral: Exercise Therapy

INTERVENTIONS:
Behavioral: Virtual Reality — Virtual Reality Based Rehabilitation including static balance, dynamic balance and walking
  Other Names: Nintendo Wii
  Arms: Virtual Reality
Behavioral: Exercise Therapy — The conventional physical Therapy program includes parameters for improving strength, flexibility, transfers, posture, balance and coordination, and sensory stimulation. These activities consist of various types of exercises that focus on lower extremity movements.
  Other Names: Conventional Physical Therapy
  Arms: Exercise Therapy

SUMMARY:
Parkinson's Disease (PD) is one of the most common neurodegenerative disease. Bradykinesia, tremor, resting tremor and postural instability are the main motor characteristics of this disease. As the disease progresses, mobility, walking, balance are reducing, the risk of falls is increasing and patients become functionally dependent. Along with these symptoms, cognitive functions are also disturbed. The most commonly distorted cognitive functions are executive functions such as planning and reasoning, working memory, episodic memory, attention and visual-spatial skills. Pharmacological and surgical treatments are used in Parkinson's disease. Pharmacologic treatment has a proven effect on motor symptoms, but since there is no approved pharmacologic treatment which has a direct effect on cognitive functions, recent studies suggest non-pharmacological treatments to improve cognitive function. Physiotherapy is also accepted among non-pharmacological treatments. Conventional physiotherapy focuses on optimizing patient independence and safety, focusing on hinting strategies, cognitive movement strategies and exercises utilizing transfers, posture, upper extremity function, balance (and falls), gait, physical capacity and (in)activity. Virtual Reality (VR) technology, a promising commonly used new rehabilitation tool, is a treatment method that can be used as one of the non-pharmacological treatment methods in Parkinson's Disease. In order to understand how neuronal network dysfunction in the Parkinson's Disease leads to clinical symptoms, both the component elements and the interconnections within these networks need to be examined in greater detail. Studies of resting state-fMRI (rs-fMRI) use correlation of activation of brain regions and time series fluctuations between brain regions to give information about connectivity in brain.

The purpose of this study is to investigate the therapeutic effects of virtual reality on motor and cognitive symptoms of PD. Furthermore, the investigation of possible effects of this effect on neuroplasticity through functional brain networks is our other objective. This study will be the first study to evaluate the plasticity effect of virtual reality application with rs-fMRI in Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* To be 50 years old and older
* Clinical diagnosis of PD within the -framework of Brain Bank criteria
* Getting a stable antiparkinsonian medication at least for the last 1 month (or the treatment has not changed)

Exclusion Criteria:

* Having a story of unstable medical condition
* History of head trauma, stroke, or exposure to toxic substances
* Implying Parkinson plus syndromes in neurological examinations; pyramidal, cerebellar examination findings, gaze paresis, autonomic dysfunction
* Being diagnosed with Dementia

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-08-18 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Motor Level | Change from Baseline at 4 weeks.
  Unified Parkinson's Disease Rating Scale-Motor (UPDRS-III)
Cognitive Level | Change from Baseline at 4 weeks.
  Montreal Cognitive Asssessment (MoCA)
Neuroplasticity | Change from Baseline at 4 weeks.
  Resting State Networks functional connectivity

SECONDARY OUTCOMES:
Balance | Change from Baseline at 4 weeks.
  Berg Balance Scale (BBS)
Quality of Life in patients with Parkinson's Disease | Change from Baseline at 4 weeks.
  The Parkinson's Disease Questionnaire (PDQ-39)
Mobility | Change from Baseline at 4 weeks.
  Timed Up and Go Test (TUG),
Functional Capacity | Change from Baseline at 4 weeks.
  Six Minute Walk Test (6MWT)
Depression | Change from Baseline at 4 weeks.
  The Geriatric Depression Scale (GDS)
Balance Confidence | Change from Baseline at 4 weeks.
  The Activities-specific Balance Confidence (ABC) Scale
Cognitive Assessment | Change from Baseline at 4 weeks.
  Neuropsychological assessment test (NPT) battery

CONTACTS AND LOCATIONS:
Overall Officials: Farzin Hajebrahimi, Principal Investigator — Medipol University; Lutfu Hanoglu, Professor, Study Director — Medipol University
Locations (1):
- Istanbul Medipol University Hospital, Istanbul, Bağcılar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be available to the public.

REFERENCES:
- [Background] Dockx K, Bekkers EM, Van den Bergh V, Ginis P, Rochester L, Hausdorff JM, Mirelman A, Nieuwboer A. Virtual reality for rehabilitation in Parkinson's disease. Cochrane Database Syst Rev. 2016 Dec 21;12(12):CD010760. doi: 10.1002/14651858.CD010760.pub2. PMID 28000926
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886